CLINICAL TRIAL: NCT05131412
Title: Mesenchymal Stem Cells for the Treatment of Pneumonia Post Haematopoietic Stem Cell Transplantation: a a Retrospective Cohort Study
Brief Title: Mesenchymal Stem Cells for the Treatment of Pneumonia Post Haematopoietic Stem Cell Transplantation
Acronym: MSCTPHSCT
Status: Completed | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xu Yang, Principal Investigator, Guangzhou Women and Children's Medical Center
Other Study IDs: GWCMC_HJ_XY_001
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Pneumonia; Hematopoietic Stem Cell Transplantation
Keywords: Mesenchymal Stromal Cell; Pneumonia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mesenchymal stromal cell: Patients treated with mesenchymal stromal cell
- non-mesenchymal stromal cell: Patients treated without mesenchymal stromal cell

SUMMARY:
The aim of this study is to determine whether mesenchymal stromal cell (MSC) treatment contribute to the good prognosis in patients with transplant-related complication, pneumonia post hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is a standard therapy strategy for most hematologic disorders and malignancies. Despite the improved survival attributed to advances in HSCT including transplantation techniques and supportive care, transplant-related pneumonia (severe pneumonia in particular) remains the leading cause of death for most HSCT patients and a major challenge for clinicians.

Mesenchymal stromal cells (MSCs), a form of multipotent cells, have been applied in therapy for various intractable disorders. MSC exerts its therapeutic effect through various biological functions including immunoregulation, tissue repairing, self-renew and differentiating into various cell lines. The American Thoracic Society has also suggested MSCs as a cell therapy agent for lung diseases. However, MSC therapy for pneumonia following HSCT has not been well investigated.

By investigating the efficacy of MSC treatment for HSCT-related pneumonia via comparing the outcomes in patients with and without MSC treatment, this study will provide a promising therapy for HSCT-related pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* patients with pneumonia after HSCT;
* patients under the age of 18 years;
* patients with normal pulmonary function before HSCT.

Exclusion Criteria:

* patients with other severe complications in progress when pneumonia occurred.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who underwent hematopoietic stem cell transplantation (HSCT) in Guangzhou Women and Children's Medical Center and got pneumonia after HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
overall cure rate | 12 months
  the proportion of cured cases in all cases
time to cure | 12 months
  the time from the first diagnosis of pneumonia to a cure was achieved

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, Study Director — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China